CLINICAL TRIAL: NCT03780738
Title: A Validation Study of The Relationship Between ALDH2 and Aortic Dissection
Acronym: VaRALAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018GDSRMvalidation
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-08

CONDITIONS: Aortic Dissection
Keywords: Aortic dissection; Aldehyde dehydrogenase 2 polymorphism
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 ml vein blood samples were collected from aortic dissection or controls in tubes containing EDTA. The samples would be centrifuged and saved in a -80℃ ultra-low temperature refrigerator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Chinese Han people to do physical examination in physical examination center of Guangdong Provincial People's Hospital
- Aortic dissection: Chinese Han people diagnosed with aortic dissection in Guangdong Provincial People's Hospital

SUMMARY:
The purpose of this study is to validate the impact of ALDH2 Glu504Lys polymorphism on aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Han people diagnosed with aortic dissection in Guangdong Provincial People's Hospital

Exclusion Criteria:

* Aortic dissection based on trauma, connective tissue diseases and pregnancy
* Patients with tumor
* Patients with no written consensus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with aortic dissection in Guangdong Provincial People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with different ALDH2 genotype | 1-30 days after samples collected
  DNA was extracted from venous blood;genomic DNA underwent PCR amplification; finally, PCR products were purified and directly sequenced by Invitrogen Corp or Biosune Corp.Then ALDH2 genotype was distinguished depend on a G-to-A missense mutation on exon 12 of ALDH2 gene.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guanzhou, Guangdong, China